CLINICAL TRIAL: NCT03413995
Title: Phase II Trial of Rucaparib in Patients With Metastatic Hormone-Sensitive Prostate Cancer Harboring Germline DNA Repair Gene Mutations (TRIUMPH)
Brief Title: Trial of Rucaparib in Patients With Metastatic Hormone-Sensitive Prostate Cancer Harboring Germline DNA Repair Gene Mutations
Acronym: TRIUMPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J17187; IRB00156514 (Other: JHMIRB)
Record Dates: First submitted 2018-01-18; First posted 2018-01-29 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer Metastatic
Keywords: metastatic hormone sensitive
MeSH Terms: interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rucaparib 600 mg BID, continuous dosing (Experimental): Rucaparib 600mg by mouth twice daily, continuous dosing
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Continuous dosing

SUMMARY:
The aim of this research is to find out if the study drug rucaparib leads to lowering of PSA levels in men with metastatic prostate cancer that has not yet been treated with androgen deprivation therapy (also referred to as metastatic hormone sensitive prostate cancer) and who have an inherited mutation in a gene involved in repairing DNA damage. The research will also examine if rucaparib is safe in individuals with metastatic prostate cancer.

Prior research studies have shown that drugs like rucaparib can be of benefit to patients with advanced metastatic prostate cancer who are resistant to androgen deprivation therapy AND who carry a mutation in a DNA repair gene. We are studying if rucaparib will be an effective treatment for these patients earlier in their treatment course (for example, prior to the start of medicines that lower testosterone level). It is unknown whether rucaparib will have the same benefit in men with metastatic prostate cancer carrying a mutation in a DNA repair gene, prior to the use of medicines that lower your testosterone level.

DETAILED DESCRIPTION:
With respect to germline mutations, a recent study found that the incidence of inherited DNA-repair gene alterations in metastatic prostate cancer to be significantly higher (11.8%) than in both men with localized prostate cancer (4.6%) and in the general population at large (2.7%). Specifically, mutations in 7 genes (ATM, BRCA1, BRCA2, CHEK2, PALB2, RAD51D, GEN1) were significantly enriched in patients with metastatic prostate cancer compared to the general population. These findings suggest that a subset of men are more likely to develop metastatic prostate cancer (i.e. those with germline mutations in DNA-repair genes) and may potentially benefit from PARPi therapy.

The clinical activity of PARPi in patients with DNA-repair mutations and metastatic prostate cancer has now been established. Focusing specifically on patients with a germline mutation in a pre-specified group of DNA-repair genes, we hypothesize that targeted therapy with PARPi should be sufficient to induce a clinical response irrespective of hormonal (castration-sensitive or castration-resistant) status. Our hypothesis is based largely on the data from Mateo et al showing a clinical response rate of 88% in a heavily pre-treated population of mCRPC patients with a DNA repair mutation, with the most pronounced responses being in men with germline inactivation.

For men with mHSPC, this trial would also provide an alternative to ADT. Identification of a non-hormonal based therapy is warranted as ADT is associated with a shorter time to castration resistance in men harboring a germline DNA repair mutation versus those with intact DNA repair. However, given that primary ADT (in mHSPC) is a standard first-line therapy, all patients on trial must be ineligible for or decline standard-of-care hormonal treatment. For patients with mHSPC who do not respond to PARPi, we will build safety rules into the trial design to take patients off study at first signs of progression. Primary ADT (mHSPC) would still remain a treatment option upon progression.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.
* Males aged 18 years of age and above
* Histological or cytologic proof of adenocarcinoma of the prostate
* Germline mutation in one or more homologous recombination DNA-repair genes (BRCA1, BRCA2, ATM, CHEK2, NBN, RAD50, RAD51C, RAD51D, PALB2, MRE11, FANCA, FANCB, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCI, FANCL, FANCM) as documented by a clinical CLIA-grade, genetic test (including but not limited to Invitae, Color Genomics, etc)
* All patients must be ineligible for or have declined androgen deprivation therapy (ADT)-based systemic treatment
* Absolute PSA ≥2.0 ng/ml at screening.
* Radiographic evidence of metastatic disease by CT scan and bone scan, performed within the prior 8 weeks.
* Serum testosterone ≥ 100 ng/dl.
* Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT))
* Participants must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

  * Estimated creatinine clearance = (140-age [years]) x weight (kg) serum creatinine (mg/dL) x 72
* ECOG Performance Status <2
* Participants must have a life expectancy ≥ 12 months.
* Male participants and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination [see appendix E for acceptable methods], throughout the period of taking study treatment and for 6 months after last dose of study drug to prevent pregnancy in a partner.

Exclusion Criteria:

* Current active second malignancy (history of non-melanoma skin cancers and superficial bladder cancers are allowed)
* Prior ADT in the past 6 months. Prior ADT in context of neoadjuvant/adjuvant primary is allowed; prior ADT for biochemical recurrence is also allowed, as long as no ADT has been administered in past 6 months and testosterone has recovered (>100 ng/dl). The total duration of prior ADT should not exceed 24 months.
* Prior oral anti-androgen (e.g. bicalutamide, nilutamide, enzalutamide, apalutamide), or androgen synthesis inhibitor (e.g. abiraterone, orteronel) in the past 6 months is not permitted. 5-alpha reductase inhibitor therapy (e.g. finasteride, dutasteride) is allowed, as long as subject has been stable on medication for past 6 months.
* Presence of visceral (i.e. lung or liver) metastases >3cm in long-axis dimension.
* Pain due to bone metastases requiring narcotic analgesics.
* Prior treatment with intravenous chemotherapy.
* Use of any prohibited concomitant medications (Appendix B: Medications With the Potential for Drug-Drug Interactions) within the prior 2 weeks.
* Involvement in the planning and/or conduct of the study (applies to both Clovis Oncology staff and/or staff at the study site)
* Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 1 month.
* Any previous treatment with a PARP inhibitor, including rucaparib.
* Resting ECG with QTc > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Major surgery within 2 weeks of starting study treatment, and patients must have recovered from any effects of any major surgery.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease, or any psychiatric disorder that prohibits obtaining informed consent.
* Unable to swallow orally administered medication or gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for HIV. Known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Known hypersensitivity to rucaparib or any of the excipients of the product.
* Whole blood transfusions in the last 30 days prior to entry to the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Markowski, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nientiedt C, Duensing A, Zschabitz S, Jager D, Hohenfellner M, Stenzinger A, Duensing S. PARP inhibition in prostate cancer. Genes Chromosomes Cancer. 2021 May;60(5):344-351. doi: 10.1002/gcc.22903. Epub 2020 Oct 28. PMID 33084183

RESULTS

PARTICIPANT FLOW:
Groups:
- Rucaparib 600 mg BID: Subjects will be administered Rucaparib 600mg by mouth twice daily, continuous dosing in 28 day cycles. Drug should be taken as close as possible to 12 hours apart and preferably at the same times every day, with water. Rucaparib tablets must be swallowed whole and may be taken with or without food.
  Rucaparib: Rucaparib will be dispensed to patients on Day 1 and every 28 days thereafter until the patient completes the study, withdraws from the study or closure of the study.
Period: Overall Study
Arm/Group | Rucaparib 600 mg BID
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rucaparib 600 mg BID, Continuous Dosing
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 68 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prostate Specific Antigen (PSA) >=50 Response
Description: Response Rate(PSA) Prostate Specific Antigen to rucaparib for patients with metastatic hormone sensitive prostate cancer harboring germline mutation in homologous recombination DNA (Deoxyribonucleic acid) repair gene. Measured by decline in PSA to 50% of baseline, confirmed with second measurement at least 4 weeks apart.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib 600 mg BID
Number analyzed (Participants) | 12
Participants | 5

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: As assessed by CTCAE v4.0
Time Frame: 4 years 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib 600 mg BID
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: PSA Progression-free Survival
Description: Defined as a time (months) from initiation of rucaparib therapy until PSA increase of 25 %, confirmed with another measurement at least 3 weeks later
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib 600 mg BID
Number analyzed (Participants) | 12
months | 11.2 [3.7 to NA] — Upper bound is not reached because there is not sufficient number of patients who have had PSA PFS events.

4. Secondary Outcome: Progression-free Survival
Description: Defined as time (months) from initiation of rucaparib therapy to radiographic or clinical progression or death, whichever comes first.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib 600 mg BID
Number analyzed (Participants) | 12
months | 12 [8.0 to NA] — Upper bound is not reached because there is not sufficient number of patients who have had PSA PFS events.

5. Secondary Outcome: Objective Response
Description: Defined as patients achieving a complete or partial response in target lesions found on radiographic scans among patients who have measurable disease at baseline.
Time Frame: 2 years
Population: Of the 12 subjects enrolled in the trial, 5 of them had measurable disease. Therefore, for this outcome, 5 were included in this outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib 600 mg BID
Number analyzed (Participants) | 5
Participants | 3

ADVERSE EVENTS:
Time Frame: Baseline to End of Treatment approximately 4 years 8 months
Arm/Group | Rucaparib 600 mg BID
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib 600 mg BID (N=12)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib 600 mg BID (N=12)
Aspartate Aminotransferase-increased (Blood and lymphatic system disorders) | 7 (7)
Alanine Aminotransferase-Increased (Blood and lymphatic system disorders) | 7 (7)
Creatinine-Increased (Blood and lymphatic system disorders) | 6 (6)
Edema (General disorders) | 1 (1) — Lower Extremity
Nausea (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 8 (8)
Dysguesia (Nervous system disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Palmar-Plantar Erythrodyesia Syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03413995/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT03413995/ICF_001.pdf